CLINICAL TRIAL: NCT03553537
Title: Multi-center Randomized Study to Compare Efficacy and Safety of Decitabine Plus CHOP (D-CHOP) Versus CHOP in Patients With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: Efficacy and Safety of Decitabine Plus CHOP vs CHOP in Patients With Untreated Peripheral T-Cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Jieping Chen, Head of Hematology Department, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-CHOP study
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell Lymphoma, decitabine
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Decitabine; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decitabine + CHOP regimen (Experimental): decitabine plus CHOP (D-CHOP) administered in 4 week cycles for 6 cycles
  Interventions: Drug: Decitabine; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- CHOP regimen (Active Comparator): cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Decitabine — 10mg/m² iv on day 1-5
  Other Names: 5-aza-2'-deoxycytidine
  Arms: Decitabine + CHOP regimen
Drug: Cyclophosphamide — 750mg/m² iv on day 6
  Other Names: CTX
Drug: Doxorubicin — DOX
  Other Names: 50mg/m² iv on day 6
Drug: Vincristine — 1.4mg/m² iv on day 6
  Other Names: VCR
Drug: Prednisone — 100mg/m² po on day6-10
  Other Names: PED

SUMMARY:
Primary objective of the study is to compare the efficacy and safety of decitabine plus CHOP (D-CHOP) versus CHOP alone in patients with previously untreated peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
This is a randomized, multi-center, open-label study to compare efficacy and safety of D-CHOP with standard CHOP regimen in patients with previously untreated PTCL. Study subjects are patients with histologically proven PTCL. Patients are randomized 1:1 to receive either cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles or decitabine plus CHOP (D-CHOP) administered in 4 week cycles for 6 cycles. In the D-CHOP arm, decitabine will be administered at a dose of 10 mg/m² IV on day 1-5 every 3 weeks. This study is divided into three phases: screening phase, treatment phase and follow-up phase. Patients will receive study drug(s) for up to 6 cycles, or until unacceptable toxicity will develop or progression or voluntary withdrawal.Adverse event of every treatment cycle will be recorded.Therapy efficacy will be evaluated after finishing 3 cycles and finishing 6 cycles therapy. Patients will be followed until disease progression, died or 2 years from the last patient randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven untreated peripheral T-cell lymphoma (include PTCL not otherwise specified, angioimmunoblastic T cell lymphoma, anapestic large cell lymphoma, enteropathy-associated T cell lymphoma, Monomorphic epitheliotropic intestinal T-cell lymphoma, Nodal peripheral T-cell lymphoma with TFH phenotype and Follicular T-cell lymphoma).
2. Males and females of 18 years of age to 80 years of age.
3. Patients have not received anti-tumor therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
5. Fit chemotherapy indications and basic requirements, including no obvious abnormal function of heart, liver, lung and kidney: creatine ≤2.0×ULN, total bilirubin ≤2.0mg/dl, transaminases≤3×ULN.
6. Normal peripheral hemogram: ANC≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^12/L.
7. None of other serious disease conflict with the therapeutic regimen.
8. None of other malignant tumor.
9. Pregnancy test of women at reproductive age must be negative.
10. Estimated survival time ≥ 3 months with good compliance.
11. Voluntary participation, cooperate with the experimental observation, and sign a written informed consent.

Exclusion Criteria:

1. Patients with the following PTCL subtypes are excluded; extranodal NNK/T-cell lymphoma, T-prolymphocytic leukemia, T large granular lymphocytic leukemia, chronic lymphoproliferative disorder of NK cells, aggressive natural killer-cell leukemia, adult T-cell leukemia/ lymphoma, hepatosplenic T-cell lymphoma, subcutaneous panniculitis-like T-cell lymphoma, cutaneous T cell lymphoma, breast implant-associated anaplastic large-cell lymphoma.
2. Transformed lymphoma.
3. Patients with other malignancies in the past or now; or secondary lymphoma triggered by chemotherapy or radiotherapy of other malignancies.
4. Already initiated lymphoma therapy (exept for the prephase treatment specified for this study).
5. Patients with primary central nervous system lymphoma or lymphoma involving central nervous system.
6. Patients who have central nervous system or meninges involvements.
7. Candidate for hematopoietic stem cell transplantation.
8. Known hypersensitivity to medications to be used.
9. Hemogram abnormality: ANC<1.5×10^9/L; or HGB<90 g/L; or PLT<100×10^9/L.
10. Known hepatic and renal insufficiency (creatine>2.0×ULN, total bilirubin>2.0 mg/dl，transaminases>3.0×ULN).
11. Patients with decompensated heart failure; or with dilated cardiomyopathy; or with coronary heart disease of non-corresponding ST-segment in ECG diagnosis; or with myocardial infarction within 6 months.
12. Patients with serious uncontroled acute infection need to be treated with antibody therapies, or antiviral therapies; or serious accompanying disorder or impaired organ function.
13. Know HIV-positivity; or HbsAg positivity; or HCV-Ab positivity.
14. Pregnancy or lactation period.
15. Patients who participated in other clinical trials within 3 months.
16. The researchers considered that patients should not be in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years
  from date of inclusion to date of progression, relapse, or death from any cause

SECONDARY OUTCOMES:
Overall Survival | 3 years
  from the date of inclusion to date of death, irrespective of cause
Response rate | 3 years
  complete response (CR) and partial response (PR) rates, using the standard response criteria (Cheson and al.)
Adverse Events | 3 years
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jieping Chen, MD,PhD, Principal Investigator — Southwest Hospital, China; Xi Li, MD, Principal Investigator — Southwest Hospital, China

IPD SHARING:
Plan to Share IPD: No